CLINICAL TRIAL: NCT02981511
Title: Assessing the Potential Use of Optiflow as a Preoxygenation Method Prior to Anaesthesia.
Brief Title: Optiflow Preoxygenation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RHMCRI0333
Record Dates: First submitted 2016-12-01; First posted 2016-12-05 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-12

CONDITIONS: Preoxygenation, Apnoea, Anaesthesia
MeSH Terms: conditions — Apnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: optiflow — Optiflow device used for preoxygenation

SUMMARY:
Optiflow can be used to prolong the apnoea period under anaesthesia without falls in blood oxygen saturation. This study is designed to assess whether the Optiflow system can efficiently replace conventional anaesthetic mask and circuit preoxygenation so that it could be used in emergency anaesthesia. If so, it would be then be in place in the case of difficult or failed intubation to maintain oxygenation ie: it could preoxygenate and then maintain oxygenation seamlessly.

DETAILED DESCRIPTION:
The Optiflow device is used to deliver high flow humidified oxygen/air via nasal cannulae to patients who have respiratory problems. More recently it has been used in patients having surgery on their larynx who are intentionally paralysed under anaesthesia where the surgeon does not want any tubes in the airway. This makes access for surgery easier/possible. Perhaps surprisingly, these patients can be left apnoeic for 30 minutes without falls in blood oxygen levels. The lungs are oxygenated despite there being no in and out breathing/ventilation.

We propose that applying Optiflow at the start of an emergency anaesthetic may be beneficial when an anaesthetist finds that tracheal intubation is impossible - a "failed intubation" scenario. Optiflow might maintain oxygenation during further attempts at intubation or until more skilled anaesthetists arrive.

Another alternative technique presently in common use is for the patient to breathe 100% oxygen via a facemask and conventional anaesthetic circuit for 3 minutes before anaesthesia starts (preoxygenation). This fills the functional residual capacity of the lungs to about 90% oxygen giving an oxygen reserve when the breathing stops until the anaesthetist breathes for them after intubating the trachea. This can result in the maintenance of normal blood oxygen saturation for several minutes longer than would be the case if the lungs had only been exposed to air before anaesthesia.

The research question that we ask is whether we can just use Optiflow instead of the conventional mask/circuit to preoxygenate patients to a similar extent and as quickly as using a facemask so that, in emergency surgery, Optiflow could be used to preoxygenate and then already be in place in case there is a failed intubation. This would enable Optiflow to be used for both purposes seamlessly without the need to switch between the two methods of oxygenation.

Research to date has not yet identified how long Optiflow needs to be in place before anaesthesia for it to be able to produce adequate preoxygenation of the lungs before the patient stops breathing. The 3 minute timing for preoxygenation is important in emergency cases e.g. when there is an emergency caesarean section to be done and every minute before the baby is delivered matters. If it were not possible to preoxygenate a patient's lungs within 3 minutes using Optiflow we would suggest that it is inappropriate to replace conventional mask pre-oxygenation and that its value in emergency anaesthesia might be reduced (although it may still have potential for less urgent anaesthesia when it could be applied for a longer duration before anaesthesia).

This will be a pilot study with 20 healthy volunteer students as subjects who will undergo an up / down sequential analysis of Optiflow pre-oxygenation. They will be recruited from posters inviting them to consider enrolling in the project. They will receive a subject information sheet and will provide written informed consent.

On the study day an individual subject will lie supine on a trolley and the Optiflow device will be fitted ready to administer humidified 100% oxygen at 45 l/min via the device's nasal cannulae. The subject will be asked to breathe normally with a closed mouth and the device will be switched on.

The initial test period will be for 3 minutes and at the end of that time the device will be turned off with the subject holding their breath in inspiration and the subject will then exhale and then breathe normally via a mouthpiece which has a side sampling port connected to a standard gas monitor (as used during anaesthesia) which will measure and display the expired oxygen percentage. This is known to equate very well to the alveolar oxygen fraction in healthy subjects and the target value will be 85%.

After the initial test the subject will be asked to walk around breathing room air for at least 15 minutes to return their lung gases to pre test normality.

The process will then be repeated as before but for a different duration:

If the target of 85% had not been reached within 3 minutes the 2nd test would be for 5 minutes.

If the 85% target had been reached the 2nd test would be reduced to 2.5 minutes.

The test runs would continue in the same up/down fashion until the minimum time required to reach 85% had been identified (to the nearest 30 seconds) or the subject had done test runs up to 10 minutes long without reaching the target.

If the subject wished to split the test runs over more than one session that would be accommodated. They would also be free to leave the study at any time if they so desired.

Subsequent subjects will have an initial test duration adjusted to the average of the previous subjects so that they may not be required to undergo as many tests (this presumes that there is not too much variation within the population) and will be less inconvenienced.

ELIGIBILITY:
Inclusion Criteria:

* healthy (ASA1or 2)

Exclusion Criteria:

* respiratory disease

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
time to end tidal oxygen content of 0.85 | less than 10 minutes
  time to this end point will be found by up/down sequential tests

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Southampton, Southampton, Hants, United Kingdom

IPD SHARING:
Plan to Share IPD: No